CLINICAL TRIAL: NCT00940615
Title: Aerobic Exercise in TBI: White Matter Integrity and Cognition
Brief Title: The Effect of Aerobic Exercise on Mild Traumatic Brain Injury
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Primary Investigator is no longer employeed by the VA
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Cox, David - Principal Investigator, Department of Veterans Affairs
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B6859-M
Record Dates: First submitted 2009-07-14; First posted 2009-07-16 (Estimated); Last update posted 2015-06-26 (Estimated); Status verified 2015-06

CONDITIONS: Traumatic Brain Injury
Keywords: traumatic brain injury; aerobic exercise; Diffusion Tensor Imaging; Neuropsychology; Rehabilitation
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): participants in the aerobic exercise intervention
  Interventions: Other: aerobic exercise
- 2 (Active Comparator): participants in the stretching/toning control condition
  Interventions: Other: stretching/toning

INTERVENTIONS:
Other: aerobic exercise — , participants assigned to the exercise treatment group of the proposed study will participate in an aerobic exercise regimen of brisk walking on a treadmill for a 60 minute interval, three times a week
  Arms: 1
Other: stretching/toning — Individuals in the control group will participate in a low intensity stretching and toning session for 60 minutes, three times a week
  Arms: 2

SUMMARY:
The current project will examine the effects of aerobic exercise on cognition among a group of veterans who have suffered a mild traumatic brain injury.

DETAILED DESCRIPTION:
There is substantial evidence that a large number of individuals who experience TBI will demonstrate life-long deficits in cognitive or social functions. An estimated 80-90,000 Americans with TBI suffer life-long impairment of physical, cognitive, and psychosocial skills to the degree that they are unable to return to school or work. Research on rehabilitation for mTBI has been minimal and typically has focused on speech, pain management, dizziness, fatigue, irritability, and sensory disorders. The results of the few studies that have examined long-term cognitive effects of mTBI have offered conflicting results. The current research will investigate the efficacy of an aerobic exercise intervention among individuals with mild traumatic brain injury (mTBI). This project will examine changes in fractional anisotropy (FA) values and cognitive functioning among individuals diagnosed with mTBI in a monitored aerobic exercise regimen, versus a low impact stretching and toning control group.

ELIGIBILITY:
Inclusion Criteria:

* Anyone between 18 and 50 years of age,
* from the geographic region served by the Malcolm Randall-North Florida-South Georgia VAMC,
* who have sustained a TBI and demonstrate impairment on neuropsychological assessment (criteria for mTBI will be defined as a loss of consciousness for not more than 30 minutes and post-trauma amnesia of not more than 24 hours).

Exclusion Criteria:

* TBI occurring less than 6 months or greater than 5 years prior to enrollment,
* any metal implants or shrapnel that may put them at risk for injury during an MRI scan,
* significant cognitive impairment (MMSE<24),
* history of stroke,
* B-12 deficiency,
* hypothyroidism,
* organ failure (renal, hepatic, cardiac, or lung),
* substance abuse,
* seizures,
* or any limitation that would preclude them from safely engaging in the aerobic exercise regimen.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2009-09; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Diffusion Tensor Imaging | 16 weeks

SECONDARY OUTCOMES:
Trail Making Test - Part A | 16 weeks
Symbol Search | 16 weeks
California Verbal Learning Test - Second Edition (CVLT-II). | 16 weeks
Brief Visual Memory Test - Revised (BVMT-R). | 16 weeks
Adaptive Digit Ordering Test (DOT-A). | 16 weeks
Continuous Performance Test of Attention (CPT-A). | 16 weeks
Delis-Kaplin Executive Function System Tower Test | 16 weeks
Trail Making Test - Part B. | 16 weeks
Controlled Oral Word Association Test (COWAT). | 16 weeks
Boston Naming Test (BNT). | 16 weeks
Judgment-Line Orientation (JLO). | 16 weeks
Grooved Pegboard Test | 16 weeks
Hand Dynamometer | 16 weeks
Finger Tapping Test | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: David E Cox, PhD, Principal Investigator — North Florida/South Georgia Veterans Health System
Locations (1):
- North Florida/South Georgia Veterans Health System, Gainesville, Florida, United States